CLINICAL TRIAL: NCT04856553
Title: Acute Effects of Handgrip on Vascular Function and Ambulatory Blood Pressure in Hypertensive Adults: A Randomized Controlled Trial
Brief Title: Acute Effects of Handgrip on Blood Pressure in Hypertensive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Aline Mendes Gerage, Professor, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ACUTE HANDGRIP 2021
Record Dates: First submitted 2021-04-14; First posted 2021-04-23 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Hypertension
Keywords: Exercise; Blood pressure; Strength training; Vascular function
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Handgrip exercise (morning) (Experimental): The handgrip exercise session will be executed with four series (two in each arm) of two minutes of isometric contraction at 30% of maximum voluntary contraction, with a one-minute interval between series in the morning.
  Interventions: Other: Acute effects of handgrip exercise
- Control (No Intervention): In the control session, the participants will remain at rest for the same period of time as in the handgrip exercise protocol.
- Handgrip exercise (afternoon) (Experimental): The handgrip exercise session will be executed with four series (two in each arm) of two minutes of isometric contraction at 30% of maximum voluntary contraction, with a one-minute interval between series in the afternoon.
  Interventions: Other: Acute effects of handgrip exercise

INTERVENTIONS:
Other: Acute effects of handgrip exercise — The participants will be randomized into three sessions, handgrip exercise in the morning, handgrip exercise in the afternoon, and control performed in the morning to analyze the acute effects of handgrip exercise on blood pressure and vascular function at different times of the day. After the morning sessions, ambulatory blood pressure will also be measured for 24 hours.
  Arms: Handgrip exercise (afternoon); Handgrip exercise (morning)

SUMMARY:
The effect of handgrip training on blood pressure reduction has been demonstrated in several studies. However, acutely, there is still divergence regarding the effects of isometric handgrip exercise on blood pressure responses, especially when it is performed at different times of the day. It is suggested that the magnitude of blood pressure reduction after a single exercise session is able to predict long-term blood pressure behavior. Thus, understanding the effects of isometric handgrip exercise, performed at different times of the day, on blood pressure in adult hypertensive individuals acutely may help to understand the effects of this type of exercise chronically.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of hypertension controlled by up to three antihypertensive medications;
2. SBP levels ≤ 180 mmHg and/or DBP ≤110 mmHg;
3. no serious heart disease;
4. no upper limb musculoskeletal injury that prevents the handgrip.

Exclusion Criteria:

1. diagnosis of other cardiovascular diseases or diabetes during the study;
2. change the class and/or dose of antihypertensive medication during the study;
3. worsening of the disease (BP > 180 or use of four or more medications).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Ambulatory Blood Pressure | 24 hours after the session
  The ambulatory blood pressure will be collected for a 24-hour period using an automatic device (Dyna-MAPA, Cardios, Brazil). The device, duly calibrated, will be connected to a cuff, in the arm of preference, for the evaluation measurements. The device will be programmed to take measurements throughout the day at 15-minute intervals and during the night every 30 minutes (between 11:00 p.m. and 7:00 a.m.). All subjects will be given forms to record possible eventualities during the use of the device.

SECONDARY OUTCOMES:
Change of clinical blood pressure from pre to post session | Before, immediately after, 15 minutes and 30 minutes after the session.
  For the measurement of clinical blood pressure, the Omron HEM 742 automatic equipment will be used. Initially, the participant will remain for 10 minutes in dorsal decubitus and then a cuff appropriate for the circumference of the participant's arm will be placed. On the right arm, consecutive measurements will be taken, one minute apart, until a difference of less than 4 mmHg between two measurements is reached. For analysis purposes, the average of the last two measurements will be used, as recommended by the 7th Brazilian Guideline on Hypertension.
Change in vascular function from pre to post session | Before, immediately after and 30 minutes after the session.
  The vascular function will be assessed using the flow-mediated dilation (FMD) technique using the LOGIQ S7 Expert ultrasound device (GE Healthcare), following the recommendations of Thijssen et al. (2019). For FMD collection, the baseline diameter of the artery will be assessed before cuff inflation for a period of at least 30 seconds. The cuff will then be inflated to 50 mmHg above the individual's systolic blood pressure for five minutes, and after this period, the cuff will be deflated and diameter measurement will be assessed for three minutes. The post-deflation diameter measurement will start 30 seconds before the cuff is released. Throughout the collection, continuous measurements of the brachial artery diameter (mm) using the Doppler function will be recorded for future analyses in percentage change.

CONTACTS AND LOCATIONS:
Overall Officials: Aline M. Gerage, Dr., Principal Investigator — Universidade Federal de Santa Catarina
Locations (1):
- Universidade Federal de Santa Catarina, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No